CLINICAL TRIAL: NCT02169726
Title: A Pilot Study to Investigate Non-Invasive Metabolic Guidance for Improving Therapeutic Ultrasound Treatment of Lower Back Muscle Injuries
Brief Title: A Pilot Study Non-Invasive Guidance for Therapeutic Ultrasound Treatment of Lower Back Muscle Injuries
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg,Ph.D.,Director, Beckman Laser Institute and Medical Clinic and Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20139473
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Injury; Muscle, Back, Lower
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Musculoskeletal injuries: Diffuse Optical Spectroscopy Imaging measure blood flow,oxygen, temperature in back muscle when they are treated with therapeutic ultrasound and can improve the treatment
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Diffuse Optical Spectroscopy Imaging measure blood flow,oxygen, temperature in back muscle when they are treated with therapeutic ultrasound and can improve the treatment

SUMMARY:
Back injuries are the most common reason people seeking for effective treatment. One of the most common treatments in sports medicine for muscular injuries is therapeutic ultrasound, which is designed to heat the injured tissue and increase the flow of blood to promote healing.

DETAILED DESCRIPTION:
Researchers at Beckman Laser institute, using a technology developed at University of California, Irvine. The device call Diffuse Optical Spectroscopy, this device developed with harmless light that can measures and detect the change of blood flow, oxygen level, temperature and muscle tissue in lower back during therapeutic ultrasound therapy treatment.

The researchers can provide information in real-time tissue change before, during, and after treatments that can determine the effectiveness of the treatment and speed up recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age,
* No back injuries, No plan treatment
* Currently diagnose with back injuries, with plan treatment of therapeutic ultrasound

Exclusion Criteria:

* Minors
* Obese
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from Univesity of California Irvine Medical Center
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Normal lower back muscle | 4 weeks
  Diffuse Optical Spectroscopy Imaging measure blood flow,oxygen, temperature in back muscle when they are treated with therapeutic ultrasound and can improve the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, Irvine, California, United States